CLINICAL TRIAL: NCT00847626
Title: A Phase 3, Double-Blind, Randomized, Factorial, Efficacy and Safety Study of TAK 491 Plus Chlorthalidone Fixed-Dose Combination in Participants With Moderate to Severe Hypertension
Brief Title: Efficacy and Safety of Azilsartan Medoxomil Combined With Chlorthalidone in Participants With Moderate to Severe Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-491CLD_302; 2008-004218-28 (EudraCT Number); U1111-1113-8735 (Registry Identifier: WHO); NCT00892645 (obsolete NCT alias)
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2012-02-07 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-01

CONDITIONS: Hypertension
Keywords: Hypertensive; Blood Pressure, High; Vascular Disease; Cardiovascular Disease; Drug Therapy
MeSH Terms: conditions — Hypertension; Vascular Diseases; Cardiovascular Diseases | interventions — azilsartan medoxomil; Chlorthalidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (11):
- Azilsartan medoxomil 20 mg/chlorthalidone 12.5 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil and chlorthalidone
- Azilsartan medoxomil 20 mg/chlorthalidone 25 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil and chlorthalidone
- Azilsartan medoxomil 40 mg/chlorthalidone 12.5 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil and chlorthalidone
- Azilsartan medoxomil 40 mg/chlorthalidone 25 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil and chlorthalidone
- Azilsartan medoxomil 80 mg/chlorthalidone 12.5 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil and chlorthalidone
- Azilsartan medoxomil 80 mg/chlorthalidone 25 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil and chlorthalidone
- Chlorthalidone 12.5 mg QD (Active Comparator)
  Interventions: Drug: Chlorthalidone
- Chlorthalidone 25 mg QD (Active Comparator)
  Interventions: Drug: Chlorthalidone
- Azilsartan medoxomil 20 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil
- Azilsartan medoxomil 40 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil
- Azilsartan medoxomil 80 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil

INTERVENTIONS:
Drug: Azilsartan medoxomil and chlorthalidone — Azilsartan medoxomil 20 mg and chlorthalidone 12.5 mg combination tablets, orally, once daily for up to 8 weeks
  Other Names: TAK-491CLD
  Arms: Azilsartan medoxomil 20 mg/chlorthalidone 12.5 mg QD
Drug: Azilsartan medoxomil and chlorthalidone — Azilsartan medoxomil 20 mg and chlorthalidone 25 mg combination tablets, orally, once daily for up to 8 weeks
  Other Names: TAK-491CLD
  Arms: Azilsartan medoxomil 20 mg/chlorthalidone 25 mg QD
Drug: Azilsartan medoxomil and chlorthalidone — Azilsartan 40 mg and chlorthalidone 12.5 mg combination tablets, orally, once daily for up to 8 weeks
  Other Names: TAK-491CLD
  Arms: Azilsartan medoxomil 40 mg/chlorthalidone 12.5 mg QD
Drug: Azilsartan medoxomil and chlorthalidone — Azilsartan medoxomil 40 mg and chlorthalidone 25 mg combination tablets, orally, once daily for up to 8 weeks
  Other Names: TAK-491CLD
  Arms: Azilsartan medoxomil 40 mg/chlorthalidone 25 mg QD
Drug: Azilsartan medoxomil and chlorthalidone — Azilsartan 80 mg and chlorthalidone 12.5 mg combination tablets, orally, once daily for up to 8 weeks
  Other Names: TAK-491CLD
  Arms: Azilsartan medoxomil 80 mg/chlorthalidone 12.5 mg QD
Drug: Azilsartan medoxomil and chlorthalidone — Azilsartan medoxomil 80 mg and chlorthalidone 25 mg combination tablets, orally, once daily for up to 8 weeks
  Other Names: TAK-491CLD
  Arms: Azilsartan medoxomil 80 mg/chlorthalidone 25 mg QD
Drug: Chlorthalidone — Azilsartan medoxomil placebo and chlorthalidone 12.5 mg combination tablets, orally, once daily for up to 8 weeks
  Arms: Chlorthalidone 12.5 mg QD
Drug: Chlorthalidone — Azilsartan medoxomil placebo and chlorthalidone 25 mg combination tablets, orally, once daily for up to 8 weeks
  Arms: Chlorthalidone 25 mg QD
Drug: Azilsartan medoxomil — Azilsartan medoxomil 20 mg and chlorthalidone placebo combination tablets, orally, once daily for up to 8 weeks
  Other Names: TAK-491CLD
  Arms: Azilsartan medoxomil 20 mg QD
Drug: Azilsartan medoxomil — Azilsartan medoxomil 40 mg and chlorthalidone placebo combination tablets, orally, once daily for up to 8 weeks
  Other Names: TAK-491CLD
  Arms: Azilsartan medoxomil 40 mg QD
Drug: Azilsartan medoxomil — Azilsartan medoxomil 80 mg and chlorthalidone placebo combination tablets, orally, once daily for up to 8 weeks
  Other Names: TAK-491CLD
  Arms: Azilsartan medoxomil 80 mg QD

SUMMARY:
The purpose of this study is to determine the efficacy and safety of azilsartan medoxomil combined with chlorthalidone, once daily (QD), in participants with moderate to severe hypertension.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), hypertension is the most common attributable cause of preventable death in developed nations, as uncontrolled hypertension greatly increases the risk of cardiovascular disease, cerebrovascular disease, and renal failure. As the population ages, the prevalence of hypertension will continue to increase if broad and effective preventive measures are not implemented. Despite the availability of antihypertensive agents, hypertension remains inadequately controlled; only about one third of patients continue to maintain control successfully.

Although most antihypertensive agents are effective at the appropriate dose, the majority have side effects that limit their use. As a class, angiotensin II receptor blockers generally are considered more tolerable than other classes of antihypertensive agents. TAK-491 (azilsartan medoxomil) is an angiotensin II receptor blocker that is being evaluated by Takeda to treat essential hypertension.

Treatments for essential hypertension commonly include use of a thiazide-like diuretic, either alone or as part of combination treatment.

This study is designed to compare the antihypertensive effect and the safety and tolerability of the azilsartan medoxomil plus chlorthalidone fixed-dose combination product (TAK 491CLD FDC) with azilsartan monotherapy and chlorthalidone monotherapy during 8 weeks of treatment.

Participants in this study will be randomized to receive one of 11 possible dosing combinations of azilsartan medoxomil , chlorthalidone and placebo over an 8 week period. The total duration of the study will be approximately 13 weeks. Participants will make 12 visits to the clinic. Each participant will also be contacted by telephone 14 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is treated with antihypertensive therapy and has a post-washout mean sitting clinic systolic blood pressure greater than or equal to 160 and less than or equal to 190 mm Hg on the day prior to randomization, or the participant has not received antihypertensive treatment within 28 days prior to Screening and has a mean sitting clinic systolic blood pressure greater than or equal to 160 and less than or equal to 190 mm Hg at the Screening Visit and on the day prior to randomization.
2. Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
3. Has clinical laboratory test results within the reference range for the testing laboratory or the investigator does not consider the results to be clinically significant.
4. Is willing to discontinue current antihypertensive medications on Day -21 or on Day -28 if on amlodipine or chlorthalidone.

Exclusion Criteria:

1. Has a mean sitting clinic diastolic blood pressure greater than 119 mm Hg on the day prior to randomization.
2. Has a baseline 24-hour ambulatory blood pressure measurement reading of insufficient quality.
3. Has works a night (third) shift (defined as 11 PM [2300] to 7 AM [0700]).
4. Has an upper arm circumference less than 24 cm or greater than 42 cm.
5. Has is noncompliant with study medication during the placebo run-in period.
6. Has secondary hypertension of any etiology.
7. Has recent history of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack.
8. Has clinically significant cardiac conduction defects.
9. Has hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease.
10. Has severe renal dysfunction or disease.
11. Has known or suspected unilateral or bilateral renal artery stenosis.
12. Has a history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug.
13. Has poorly controlled type 1 or type 2 diabetes mellitus at Screening.
14. Has hypokalemia or hyperkalemia.
15. Has an alanine aminotransferase or aspartate aminotransferase level of greater than 2.5 times the upper limit of normal, active liver disease, or jaundice.
16. Has any other known serious disease or condition that would compromise safety, might affect life expectancy, or make it difficult to successfully manage and follow Has according to the protocol.
17. Has known hypersensitivity to angiotensin II receptor blockers, thiazide-type diuretics or other sulfonamide-derived compounds.
18. Has been randomized in a previous azilsartan medoxomil study.
19. Is currently participating in another investigational study or is receiving or has received any investigational compound within 30 days prior to Screening.
20. Has a history of drug abuse or a history of alcohol abuse within the past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1711 (Actual)
Dates: Start 2009-01; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Takeda
Locations (99):
- United States (84):
  - Birmingham, Alabama
  - Columbiana, Alabama
  - Tuscaloosa, Alabama
  - Chandler, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Buena Park, California
  - Carmichael, California
  - Costa Mesa, California
  - Irvine, California
  - Palm Springs, California
  - Riverside, California
  - Sacramento, California
  - San Diego, California
  - Vista, California
  - Walnut Creek, California
  - Middletown, Delaware
  - Bradenton, Florida
  - Deerfield Beach, Florida
  - Fort Lauderdale, Florida
  - Hallandale, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Longwood, Florida
  - Miami, Florida
  - Ocala, Florida
  - Ormond Beach, Florida
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Buffalo Grove, Illinois
  - Libertyville, Illinois
  - Melrose Park, Illinois
  - Fishers, Indiana
  - Indianapolis, Indiana
  - Erlanger, Kentucky
  - Madisonville, Kentucky
  - Paducah, Kentucky
  - Rockville, Maryland
  - Ann Arbor, Michigan
  - Chesterfield, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - Henderson, Nevada
  - Brick, New Jersey
  - Margate City, New Jersey
  - Albuquerque, New Mexico
  - Endwell, New York
  - Cary, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Lyndhurst, Ohio
  - Willoughby Hills, Ohio
  - Oklahoma City, Oklahoma
  - Ashland, Oregon
  - Altoona, Pennsylvania
  - Bensalem, Pennsylvania
  - Feasterville, Pennsylvania
  - Jenkintown, Pennsylvania
  - Sellersville, Pennsylvania
  - Warminster, Pennsylvania
  - Charleston, South Carolina
  - Florence, South Carolina
  - Murrells Inlet, South Carolina
  - Simpsonville, South Carolina
  - Spartanburg, South Carolina
  - Clarksville, Tennessee
  - New Tazewell, Tennessee
  - Austin, Texas
  - Bellaire, Texas
  - Dallas, Texas
  - Houston, Texas
  - McKinney, Texas
  - Richardson, Texas
  - San Antonio, Texas
  - Magna, Utah
  - West Jordan, Utah
  - Arlington, Virginia
  - Virginia Beach, Virginia
  - Oregon, Wisconsin
- Chile (2):
  - Santiago
  - Temuco
- Mexico (3):
  - Aguascalientes
  - Mexico City
  - Mérida
- Peru (8):
  - Bellavista
  - Chiclayo
  - Jesus Maria
  - Miraflores
  - San Borja
  - San Martín de Porres
  - Trujillo
  - Umacollo
- Russia (2):
  - Moscow
  - Saint Petersburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 175 investigative sites in Austria, Chile, Germany, Guatemala, Mexico, Netherlands, Peru, Poland, Russian Federation and the United States from 29 January 2009 to 10 July 2010.
Pre-assignment Details: Participants with moderate to severe essential hypertension were enrolled in one of 11, once-daily (QD) treatment groups.
Groups:
- Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD: Azilsartan medoxomil 20 mg and chlorthalidone 12.5 mg combination tablets, orally, once daily for up to 8 weeks.
- Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD: Azilsartan medoxomil 20 mg and chlorthalidone 25 mg combination tablets, orally, once daily for up to 8 weeks.
- Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD: Azilsartan 40 mg and chlorthalidone 12.5 mg combination tablets, orally, once daily for up to 8 weeks.
- Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD: Azilsartan medoxomil 40 mg and chlorthalidone 25 mg combination tablets, orally, once daily for up to 8 weeks.
- Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD: Azilsartan 80 mg and chlorthalidone 12.5 mg combination tablets, orally, once daily for up to 8 weeks.
- Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD: Azilsartan medoxomil 80 mg and chlorthalidone 25 mg combination tablets, orally, once daily for up to 8 weeks.
- Chlorthalidone 12.5 mg QD: Azilsartan medoxomil placebo and chlorthalidone 12.5 mg combination tablets, orally, once daily for up to 8 weeks.
- Chlorthalidone 25 mg QD: Azilsartan medoxomil placebo and chlorthalidone 25 mg combination tablets, orally, once daily for up to 8 weeks.
- Azilsartan Medoxomil 20 mg QD: Azilsartan medoxomil 20 mg and chlorthalidone placebo combination tablets, orally, once daily for up to 8 weeks.
- Azilsartan Medoxomil 40 mg QD: Azilsartan medoxomil 40 mg and chlorthalidone placebo combination tablets, orally, once daily for up to 8 weeks.
- Azilsartan Medoxomil 80 mg QD: Azilsartan medoxomil 80 mg and chlorthalidone placebo combination tablets, orally, once daily for up to 8 weeks.
Period: Overall Study
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Started | 156 | 154 | 147 (Includes participant who was randomized but did not receive study medication.) | 156 | 153 | 162 (Includes participant who was randomized but did not receive study medication.) | 157 (Includes participant who was randomized but did not receive study medication.) | 160 (Includes participant who was treated with double-blind study medication but not randomized.) | 155 | 153 | 162
Completed | 135 | 131 | 131 | 125 | 125 | 125 | 135 | 141 | 141 | 139 | 142
Not Completed | 21 | 23 | 16 | 31 | 28 | 37 | 22 | 19 | 14 | 14 | 20
Not completed — Adverse Event | 10 | 10 | 6 | 19 | 11 | 22 | 4 | 6 | 3 | 6 | 6
Not completed — Protocol Violation | 2 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1 | 0 | 3 | 1 | 3 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 5 | 3 | 8 | 12 | 9 | 8 | 4 | 4 | 5 | 2
Not completed — Lack of Efficacy | 3 | 1 | 0 | 1 | 2 | 0 | 6 | 2 | 5 | 1 | 7
Not completed — Other | 1 | 5 | 4 | 1 | 2 | 2 | 2 | 3 | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Total
Number analyzed (Participants) | 156 | 154 | 147 | 156 | 153 | 162 | 157 | 159 | 155 | 153 | 162 | 1714
Age Continuous [Mean (Standard Deviation); unit: years] | 58.2 (10.57) | 57.4 (11.13) | 56.2 (10.50) | 57.4 (11.07) | 55.8 (11.22) | 57.6 (11.04) | 57.3 (11.30) | 56.2 (10.04) | 57.3 (11.04) | 57.8 (10.28) | 57.3 (10.87) | 57.2 (10.82)
Age, Customized [Number; unit: participants]
  <45 years | 15 | 16 | 17 | 21 | 25 | 19 | 21 | 18 | 18 | 17 | 16 | 203
  Between 45 to 64 years | 98 | 97 | 100 | 93 | 90 | 104 | 97 | 108 | 97 | 98 | 107 | 1089
  ≥65 years | 43 | 41 | 30 | 42 | 38 | 39 | 39 | 33 | 40 | 38 | 39 | 422
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 77 | 76 | 85 | 82 | 100 | 74 | 90 | 87 | 68 | 84 | 909
  Male | 70 | 77 | 71 | 71 | 71 | 62 | 83 | 69 | 68 | 85 | 78 | 805
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 19 | 11 | 15 | 19 | 15 | 17 | 19 | 20 | 17 | 15 | 177
  Not Hispanic or Latino | 90 | 75 | 76 | 85 | 71 | 87 | 84 | 86 | 77 | 80 | 86 | 897
  Unknown or Not Reported | 56 | 60 | 60 | 56 | 63 | 60 | 56 | 54 | 58 | 56 | 61 | 640
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 9 | 13 | 13 | 13 | 12 | 16 | 14 | 14 | 11 | 13 | 14 | 142
  Asian | 4 | 3 | 4 | 4 | 2 | 3 | 1 | 7 | 1 | 1 | 4 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Black or African American | 34 | 28 | 29 | 30 | 26 | 34 | 31 | 29 | 31 | 35 | 35 | 342
  White | 111 | 112 | 102 | 111 | 114 | 109 | 111 | 111 | 113 | 105 | 111 | 1210
  More than one race | 2 | 2 | 1 | 2 | 1 | 0 | 1 | 2 | 1 | 1 | 2 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Chile | 3 | 3 | 3 | 2 | 2 | 3 | 2 | 1 | 2 | 3 | 2 | 26
  Germany | 4 | 6 | 6 | 5 | 6 | 5 | 4 | 5 | 3 | 4 | 5 | 53
  Guatemala | 8 | 8 | 9 | 10 | 10 | 8 | 8 | 9 | 8 | 9 | 9 | 96
  Mexico | 10 | 11 | 11 | 9 | 12 | 11 | 11 | 8 | 13 | 11 | 12 | 119
  Netherlands | 6 | 7 | 6 | 5 | 7 | 5 | 6 | 6 | 6 | 6 | 7 | 67
  Peru | 11 | 12 | 13 | 12 | 12 | 14 | 12 | 11 | 13 | 12 | 12 | 134
  Poland | 8 | 8 | 7 | 8 | 8 | 8 | 7 | 8 | 8 | 7 | 8 | 85
  Russian Federation | 5 | 5 | 5 | 5 | 5 | 6 | 6 | 6 | 5 | 4 | 6 | 58
  United States | 100 | 94 | 87 | 100 | 90 | 102 | 101 | 105 | 97 | 97 | 101 | 1074
Height [Mean (Standard Deviation); unit: cm] | 166.3 (11.71) | 166.6 (10.85) | 167.1 (11.44) | 166.8 (11.64) | 166.6 (10.81) | 165.4 (10.79) | 168.3 (11.07) | 166.1 (11.36) | 166.4 (10.65) | 167.7 (12.27) | 167.1 (11.85) | 166.8 (11.32)
Weight [Mean (Standard Deviation); unit: kg] | 89.85 (22.076) | 86.06 (18.056) | 89.28 (21.484) | 90.16 (21.949) | 87.31 (19.209) | 86.44 (20.412) | 89.12 (21.049) | 86.70 (20.270) | 87.27 (18.934) | 87.54 (19.019) | 86.27 (20.354) | 87.80 (20.289)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.2 (5.73) | 31.0 (5.65) | 31.8 (6.57) | 32.2 (6.01) | 31.4 (5.84) | 31.5 (6.28) | 31.2 (5.85) | 31.2 (5.78) | 31.3 (5.23) | 31.0 (5.85) | 30.8 (6.28) | 31.4 (5.92)
Smoking Status [Number; unit: participants]
  Never smoked | 94 | 84 | 81 | 79 | 91 | 94 | 93 | 91 | 92 | 90 | 94 | 983
  Current smoker | 22 | 28 | 25 | 35 | 26 | 28 | 25 | 29 | 25 | 31 | 29 | 303
  Ex-smoker | 40 | 42 | 41 | 42 | 36 | 40 | 39 | 39 | 38 | 32 | 39 | 428
Estimated glomerular filtration rate (eGFR) [Number; unit: participants] — eGFR based on calculated creatinine clearance.
  Categories:
  Normal renal function (≥90 mL/min/1.73 m2) Mild renal impairment(60 to <90 mL/min/1.73 m2) Moderate renal impairment (30 to <60 mL/min/1.73 m2) Severe renal impairment (0 to <30 mL/min/1.73 m2)
  Includes all randomized participants
  participants
    ≥0 and <30 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    ≥30 and <60 | 13 | 14 | 6 | 8 | 6 | 10 | 12 | 9 | 11 | 11 | 8 | 108
    ≥60 and <90 | 95 | 90 | 93 | 97 | 109 | 110 | 101 | 100 | 94 | 95 | 99 | 1083
    ≥90 | 48 | 50 | 48 | 51 | 38 | 42 | 44 | 50 | 49 | 46 | 55 | 521
    Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in Trough, Systolic Blood Pressure as Measured by Ambulatory Blood Pressure Monitoring (Pooled Analysis)
Description: The change in trough systolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 8.
Population: Full analysis set, defined as all randomized participants who received at least 1 dose of double-blind study medication, with both a baseline value and at least 1 post-baseline value, with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Groups:
- Azilsartan Medoxomil 40 mg or 80 mg/Chlorthalidone 25 mg QD: Azilsartan medoxomil 40 mg and chlorthalidone 25 mg combination tablets, orally, once daily for up to 8 weeks.
  OR
  Azilsartan medoxomil 80 mg and chlorthalidone 25 mg combination tablets, orally, once daily for up to 8 weeks.
Arm/Group | Azilsartan Medoxomil 40 mg or 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 228 | 134 | 127
mmHg | -28.9 (0.89) | -15.9 (1.16) | -15.1 (1.19)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg or 80 mg/Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Analysis of covariance model (ANCOVA) using treatment as a fixed effect and baseline as a covariate was performed. Results for Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD and Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD pool were obtained using contrast with coefficients of 0.5 for Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD and 0.5 for Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD from the ANCOVA model; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Net) = -13.0, 95% CI 2-sided [-15.8 to -9.5]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg or 80 mg/Chlorthalidone 25 mg QD vs Azilsartan Medoxomil 80 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed. Results for Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD and Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD pool were obtained using contrast with coefficients of 0.5 for Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD and 0.5 for Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD from the ANCOVA model; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -13.8, 95% CI 2-sided [-16.7 to -10.9]

2. Secondary Outcome: Change From Baseline to Week 8 in Trough, Sitting, Clinic Systolic Blood Pressure
Description: The change in trough systolic blood pressure measured at final visit or week 8 relative to baseline. Systolic blood pressure is the arithmetic mean of the 3 serial trough sitting systolic blood pressure measurements.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 154 | 153 | 145 | 155 | 151 | 158 | 155 | 156 | 155 | 152 | 162
mmHg | -33.8 (1.26) | -37.0 (1.26) | -36.8 (1.30) | -39.5 (1.25) | -36.9 (1.27) | -40.1 (1.24) | -21.1 (1.25) | -27.1 (1.25) | -19.8 (1.26) | -23.3 (1.27) | -24.2 (1.23)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD vs Chlorthalidone 12.5 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -12.7, 95% CI 2-sided [-16.2 to -9.2]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -9.9, 95% CI 2-sided [-13.4 to -6.4]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD vs Chlorthalidone 12.5 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -15.7, 95% CI 2-sided [-19.2 to -12.1]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -12.4, 95% CI 2-sided [-15.8 to -8.9]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD vs Chlorthalidone 12.5 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -15.8, 95% CI 2-sided [-19.3 to -12.3]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -13.0, 95% CI 2-sided [-16.5 to -9.5]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD vs Azilsartan Medoxomil 20 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -14.0, 95% CI 2-sided [-17.5 to -10.5]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD vs Azilsartan Medoxomil 20 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -17.2, 95% CI 2-sided [-20.6 to -13.7]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD vs Azilsartan Medoxomil 40 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -13.5, 95% CI 2-sided [-17.0 to -9.9]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD vs Azilsartan Medoxomil 40 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -16.2, 95% CI 2-sided [-19.7 to -12.7]
Statistical Analysis 11: Comparison: Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD vs Azilsartan Medoxomil 80 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -12.8, 95% CI 2-sided [-16.3 to -9.3]
Statistical Analysis 12: Comparison: Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD vs Azilsartan Medoxomil 80 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -16.0, 95% CI 2-sided [-19.4 to -12.6]

3. Secondary Outcome: Change From Baseline to Week 8 in Trough Systolic Blood Pressure as Measured by Ambulatory Blood Pressure Monitoring in Black Participants (Pooled Analysis)
Description: The change in trough systolic blood pressure in black subjects measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg or 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 40 | 22 | 28
mmHg | -28.2 (2.49) | -23.4 (3.36) | -9.9 (2.97)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg or 80 mg/Chlorthalidone 25 mg QD vs Azilsartan Medoxomil 80 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed. Results for Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD and Azilsartan Medoxomil 80mg/Chlorthalidone 25 mg QD pool were obtained using contrast with coefficients of 0.5 for Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD and 0.5 for Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD from the ANCOVA model; Test type: Superiority or Other; p = 0.255, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -4.8, 95% CI 2-sided [-13.0 to 3.5]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg or 80 mg/Chlorthalidone 25 mg QD vs Azilsartan Medoxomil 80 mg QD; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -18.2, 95% CI 2-sided [-25.9 to -10.6]

4. Secondary Outcome: Change From Baseline to Week 8 in Trough Systolic Blood Pressure as Measured by Ambulatory Blood Pressure Monitoring in Black Participants (Pairwise Analysis)
Description: The change in trough systolic blood pressure in black participants as measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 24 | 22 | 24 | 19 | 18 | 21 | 24 | 22 | 26 | 27 | 28
mmHg | -27.2 (3.21) | -25.4 (3.36) | -21.5 (3.21) | -31.9 (3.61) | -24.8 (3.71) | -24.4 (3.43) | -12.2 (3.22) | -23.4 (3.36) | -10.7 (3.10) | -11.0 (3.04) | -9.9 (2.97)

5. Secondary Outcome: Change From Baseline to Week 8 in Trough, Sitting, Clinic Diastolic Blood Pressure
Description: The change in trough diastolic blood pressure measured at final visit or week 8 relative to baseline. Diastolic blood pressure is the average of the 3 serial trough clinic sitting diastolic blood pressure measurements.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 154 | 153 | 145 | 155 | 151 | 158 | 155 | 156 | 155 | 152 | 162
mmHg | -14.4 (0.72) | -15.5 (0.72) | -15.6 (0.74) | -17.0 (0.72) | -16.9 (0.73) | -18.5 (0.71) | -7.4 (0.72) | -9.2 (0.72) | -6.7 (0.72) | -9.2 (0.73) | -9.9 (0.70)

6. Secondary Outcome: Change From Baseline to Week 8 in the Mean Trough Diastolic Blood Pressure (22 to 24 Hours After Dosing), as Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough diastolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 127 | 118 | 117 | 114 | 110 | 114 | 130 | 134 | 128 | 131 | 127
mmHg | -13.3 (0.80) | -15.0 (0.83) | -13.5 (0.83) | -17.3 (0.85) | -16.5 (0.86) | -16.1 (0.85) | -6.5 (0.79) | -7.5 (0.78) | -7.9 (0.80) | -7.3 (0.79) | -8.9 (0.80)

7. Secondary Outcome: Change From Baseline to Week 8 in the 24-hour Mean Systolic Blood Pressure, as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in 24-hour mean systolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 127 | 118 | 117 | 114 | 110 | 114 | 130 | 134 | 128 | 131 | 127
mmHg | -24.0 (0.97) | -26.7 (1.01) | -26.1 (1.01) | -30.4 (1.03) | -27.9 (1.04) | -28.1 (1.03) | -10.9 (0.96) | -14.7 (0.95) | -11.7 (0.97) | -12.6 (0.96) | -15.3 (0.97)

8. Secondary Outcome: Change From Baseline to Week 8 in the 24-hour Mean Diastolic Blood Pressure, as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in 24-hour mean diastolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 127 | 118 | 117 | 114 | 110 | 114 | 130 | 134 | 128 | 131 | 127
mmHg | -13.5 (0.60) | -15.0 (0.62) | -14.9 (0.63) | -17.3 (0.64) | -16.5 (0.65) | -15.9 (0.64) | -5.6 (0.59) | -6.7 (0.59) | -6.8 (0.60) | -7.6 (0.59) | -8.8 (0.60)

9. Secondary Outcome: Change From Baseline to Week 8 in the Mean Daytime (6 AM to 10 PM) Systolic Blood Pressure, as Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean systolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 127 | 118 | 117 | 114 | 110 | 114 | 130 | 134 | 128 | 131 | 127
mmHg | -24.4 (1.01) | -27.7 (1.05) | -26.7 (1.06) | -31.2 (1.07) | -28.4 (1.09) | -28.5 (1.07) | -10.8 (1.00) | -14.7 (0.99) | -11.7 (1.01) | -12.8 (1.00) | -15.7 (1.01)

10. Secondary Outcome: Change From Baseline to Week 8 in the Mean Daytime (6 AM to 10 PM) Diastolic Blood Pressure, as Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean diastolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 127 | 118 | 117 | 114 | 110 | 114 | 130 | 134 | 128 | 131 | 127
mmHg | -13.7 (0.64) | -15.6 (0.66) | -15.1 (0.66) | -17.6 (0.67) | -16.8 (0.69) | -16.2 (0.67) | -5.6 (0.63) | -6.5 (0.62) | -6.8 (0.64) | -7.7 (0.63) | -9.1 (0.64)

11. Secondary Outcome: Change From Baseline to Week 8 in the Mean Nighttime (12 AM to 6 AM) Systolic Blood Pressure, as Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean systolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 127 | 118 | 117 | 114 | 110 | 114 | 130 | 134 | 128 | 131 | 127
mmHg | -22.5 (1.09) | -24.0 (1.13) | -24.3 (1.14) | -28.1 (1.15) | -26.5 (1.17) | -26.3 (1.15) | -11.3 (1.08) | -14.4 (1.06) | -11.8 (1.09) | -11.8 (1.08) | -14.2 (1.09)

12. Secondary Outcome: Change From Baseline to Week 8 in the Mean Nighttime (12 AM to 6 AM) Diastolic Blood Pressure, as Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean diastolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 127 | 118 | 117 | 114 | 110 | 114 | 130 | 134 | 128 | 131 | 127
mmHg | -12.8 (0.71) | -13.5 (0.73) | -14.4 (0.74) | -16.2 (0.75) | -15.8 (0.76) | -14.9 (0.75) | -6.0 (0.70) | -7.1 (0.69) | -6.9 (0.70) | -7.5 (0.69) | -8.0 (0.71)

13. Secondary Outcome: Change From Baseline to Week 8 in the Mean Systolic Blood Pressure at 0 to 12 Hours After Dosing, as Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 12-hour mean systolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 127 | 118 | 117 | 114 | 110 | 114 | 130 | 134 | 128 | 131 | 127
mmHg | -24.6 (1.07) | -28.0 (1.11) | -27.1 (1.12) | -31.7 (1.13) | -28.5 (1.15) | -28.7 (1.13) | -10.4 (1.06) | -14.5 (1.04) | -11.8 (1.07) | -12.7 (1.05) | -15.8 (1.07)

14. Secondary Outcome: Change From Baseline to Week 8 in the Mean Diastolic Blood Pressure at 0 to 12 Hours After Dosing, as Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 12-hour mean diastolic blood pressure measured at final visit or week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 127 | 118 | 117 | 114 | 110 | 114 | 130 | 134 | 128 | 131 | 127
mmHg | -13.6 (0.68) | -15.6 (0.71) | -15.4 (0.71) | -17.8 (0.72) | -16.8 (0.73) | -16.2 (0.72) | -5.3 (0.67) | -6.3 (0.66) | -6.8 (0.68) | -7.6 (0.67) | -9.2 (0.68)

15. Secondary Outcome: Percentage of Participants Who Achieve a Clinic Systolic Blood Pressure Response at Week 8, as Defined by Clinic Systolic Blood Pressure <140 mm Hg and/or a Reduction of ≥20 mm Hg From Baseline.
Description: Percentage of participants who achieve a clinic systolic blood pressure response measured at week 8, defined as less than 140 mm Hg and/or reduction from baseline of greater than or equal to 20 mm Hg. Systolic blood pressure is the average of the 3 serial trough sitting clinic systolic blood pressure measurements.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 154 | 153 | 145 | 155 | 151 | 158 | 155 | 156 | 155 | 152 | 162
percentage of participants | 86.4 | 88.9 | 90.3 | 93.5 | 86.8 | 94.9 | 56.1 | 76.9 | 53.5 | 64.5 | 66.7

16. Primary Outcome: Change From Baseline to Week 8 in Trough, Systolic Blood Pressure as Measured by Ambulatory Blood Pressure Monitoring (Pairwise Analysis)
Description: as for outcome 1
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 127 | 118 | 117 | 114 | 110 | 114 | 130 | 134 | 128 | 131 | 127
mmHg | -22.9 (1.19) | -26.3 (1.24) | -24.4 (1.24) | -29.8 (1.26) | -26.3 (1.28) | -28.0 (1.26) | -12.7 (1.18) | -15.9 (1.16) | -12.1 (1.19) | -12.8 (1.17) | -15.1 (1.19)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD vs Chlorthalidone 12.5 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -10.3, 95% CI 2-sided [-13.6 to -7.0]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -10.4, 95% CI 2-sided [-13.7 to -7.0]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD vs Chlorthalidone 12.5 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -11.8, 95% CI 2-sided [-15.1 to -8.4]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -13.9, 95% CI 2-sided [-17.3 to -10.6]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD vs Chlorthalidone 12.5 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -13.7, 95% CI 2-sided [-17.1 to -10.3]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -12.0, 95% CI 2-sided [-15.4 to -8.7]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD vs Azilsartan Medoxomil 20 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -10.9, 95% CI 2-sided [-14.2 to -7.6]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD vs Azilsartan Medoxomil 20 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -14.2, 95% CI 2-sided [-17.6 to -10.9]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD vs Azilsartan Medoxomil 40 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -11.6, 95% CI 2-sided [-15.0 to -8.3]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD vs Azilsartan Medoxomil 40 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -17.0, 95% CI 2-sided [-20.4 to -13.6]
Statistical Analysis 11: Comparison: Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD vs Azilsartan Medoxomil 80 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -11.2, 95% CI 2-sided [-14.7 to -7.8]
Statistical Analysis 12: Comparison: Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD vs Azilsartan Medoxomil 80 mg QD; ANCOVA using treatment as a fixed effect and baseline as a covariate was performed; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -12.8, 95% CI 2-sided [-16.2 to -9.4]

17. Secondary Outcome: Percentage of Participants Who Achieve a Clinic Diastolic Blood Pressure Response at Week 8, Defined as Clinic Diastolic Blood Pressure <90 mm Hg and/or a Reduction of ≥10 mm Hg From Baseline.
Description: Percentage of participants who achieve a clinic diastolic blood pressure response measured at week 8, defined as less than 90 mm Hg and/or reduction from baseline of greater than or equal to 10 mm Hg. Diastolic blood pressure is the average of the 3 serial trough sitting clinic diastolic blood pressure measurements.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 154 | 153 | 145 | 155 | 151 | 158 | 155 | 156 | 155 | 152 | 162
percentage of participants | 89.6 | 89.5 | 87.6 | 94.8 | 90.1 | 96.8 | 63.9 | 78.8 | 60.6 | 71.1 | 74.7

18. Secondary Outcome: Percentage of Participants Who Achieve Both a Clinic Systolic and Diastolic Blood Pressure Response at Week 8.
Description: Percentage of participants who achieve both a clinic systolic and diastolic blood pressure response measured at week 8, defined as systolic blood pressure less than 140 mm Hg and/or reduction from baseline of greater than or equal to 20 mm Hg AND diastolic blood pressure less than 90 mm Hg and/or reduction from baseline of greater than or equal to 10 mm Hg . Systolic/diastolic blood pressure is based on the average of the 3 serial trough clinic sitting systolic/diastolic blood pressure measurements.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Number analyzed (Participants) | 154 | 153 | 145 | 155 | 151 | 158 | 155 | 156 | 155 | 152 | 162
percentage of participants | 83.1 | 84.3 | 84.8 | 91.0 | 82.8 | 93.0 | 45.8 | 67.9 | 39.4 | 55.3 | 62.3

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started on or after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD | Chlorthalidone 12.5 mg QD | Chlorthalidone 25 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD
Serious Adverse Events (participants affected / at risk) | 3/156 | 0/154 | 1/146 | 2/156 | 2/153 | 2/161 | 0/156 | 2/160 | 2/155 | 2/153 | 3/162
Other Adverse Events (participants affected / at risk) | 52/156 | 55/154 | 40/146 | 74/156 | 52/153 | 67/161 | 51/156 | 53/160 | 25/155 | 36/153 | 32/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD (N=156) | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD (N=154) | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD (N=146) | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD (N=156) | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD (N=153) | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD (N=161) | Chlorthalidone 12.5 mg QD (N=156) | Chlorthalidone 25 mg QD (N=160) | Azilsartan Medoxomil 20 mg QD (N=155) | Azilsartan Medoxomil 40 mg QD (N=153) | Azilsartan Medoxomil 80 mg QD (N=162)
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drop attacks (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radicular syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 20 mg/Chlorthalidone 12.5 mg QD (N=156) | Azilsartan Medoxomil 20 mg/Chlorthalidone 25 mg QD (N=154) | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD (N=146) | Azilsartan Medoxomil 40 mg/Chlorthalidone 25 mg QD (N=156) | Azilsartan Medoxomil 80 mg/Chlorthalidone 12.5 mg QD (N=153) | Azilsartan Medoxomil 80 mg/Chlorthalidone 25 mg QD (N=161) | Chlorthalidone 12.5 mg QD (N=156) | Chlorthalidone 25 mg QD (N=160) | Azilsartan Medoxomil 20 mg QD (N=155) | Azilsartan Medoxomil 40 mg QD (N=153) | Azilsartan Medoxomil 80 mg QD (N=162)
Nasopharyngitis (Infections and infestations) | 8 | 5 | 2 | 7 | 2 | 3 | 6 | 4 | 2 | 7 | 2
Blood creatinine increased (Investigations) | 15 | 19 | 17 | 29 | 18 | 32 | 5 | 9 | 4 | 5 | 6
Blood creatine phosphokinase increased (Investigations) | 3 | 4 | 3 | 10 | 3 | 3 | 6 | 7 | 6 | 7 | 6
Blood uric acid increased (Investigations) | 3 | 9 | 6 | 7 | 9 | 3 | 6 | 5 | 1 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 5 | 0 | 2 | 4 | 19 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 12 | 17 | 20 | 21 | 19 | 19 | 6 | 5 | 2 | 7 | 6
Headache (Nervous system disorders) | 8 | 12 | 1 | 9 | 11 | 11 | 19 | 17 | 13 | 11 | 12
Blood urea increased (Investigations) | 1 | 6 | 4 | 8 | 6 | 9 | 0 | 4 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 6 | 4 | 3 | 3 | 10 | 3 | 3 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 2 | 0 | 6 | 2 | 4 | 2 | 0 | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.